CLINICAL TRIAL: NCT01964963
Title: Alogliptin (Nesina) Tablets Special Drug Use Surveillance: Mild Type 2 Diabetes Mellitus
Brief Title: Alogliptin Tablets Special Drug Use Surveillance: Mild Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 121-015; JapicCTI-132283 (Registry Identifier: JapicCTI (Japan))
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alogliptin: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months. Participants will receive interventions as part of routine medical care.
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: Nesina; SYR-322

SUMMARY:
The purpose of this study is to examine the safety and efficacy of long-term treatment with alogliptin (Nesina) in patients with mild type 2 diabetes mellitus in the routine clinical setting.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of alogliptin, designed to investigate the safety and efficacy of treatment with alogliptin in patients with mild type 2 diabetes mellitus in the routine clinical setting.

Participants will be patients with mild type 2 diabetes mellitus. The planned sample size is 20,000.

The usual adult dosage for oral use is 1 alogliptin tablet (25 mg of alogliptin) once daily.

ELIGIBILITY:
Inclusion Criteria:

-Patients with Haemoglobin A1c (HbA1c) [Japan Diabetes Society (JDS) value] ≤7.0% at the time of enrolment (within 3 months before initiation of alogliptin therapy), regardless of the use of antidiabetic medication.

Exclusion Criteria:

-Patients contraindicated for alogliptin.

1. Patients with severe ketosis, diabetic coma or precoma, or type 1 diabetes mellitus.
2. Patients with severe infection, pre- or post-operative patients, or patients with serious traumatic injury.
3. Patients with a history of hypersensitivity to any ingredient of alogliptin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with mild type 2 diabetes mellitus who have been examined at a medical institution
Sampling Method: Non-Probability Sample
Enrollment: 19192 (Actual)
Dates: Start 2011-08-03 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1406 investigative sites in Japan, from 03 August 2011 to 31 July 2017.
Pre-assignment Details: Participants with a historical diagnosis of mild type 2 diabetes mellitus were enrolled. Participants received interventions as part of routine medical care.
Groups:
- Alogliptin 25 mg: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Alogliptin 25 mg
Started | 19192
Completed | 18249
Not Completed | 943
Not completed — Case Report Forms Uncollected | 888
Not completed — Protocol Deviation | 50
Not completed — Data Reliability was not Assured | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Arm/Group | Alogliptin 25 mg
Number analyzed (Participants) | 18249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7970
  Male | 10279
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 18249
Number of Females who were not Pregnant [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    number analyzed (Participants) | 7970
    (all) | 7970
Duration of Diagnosis of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 13939
    (all) | 6.03 (6.452)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 15139
    (all) | 159.6 (9.61)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 13073
    (all) | 63.85 (13.324)
BMI [Mean (Standard Deviation); unit: kg/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/meter (m)^2
    number analyzed (Participants) | 12378
    (all) | 24.95 (4.067)
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 18069
    Inpatient | 180
Degree of Renal Dysfunction [Count of Participants; unit: Participants] — Degree of renal dysfunction was determined by investigator for each participant.
  Participants
    Normal | 14808
    Mild | 2766
    Moderate | 598
    Severe | 77
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Presence of Medical Complications | 2322
    Had Presence of Medical Complications | 15927
Concomitant Diabetes Mellitus [Count of Participants; unit: Participants]
  Had No Concomitant Diabetes Mellitus | 16165
  Had Concomitant Diabetes Mellitus | 2084
Concomitant Hypertension [Count of Participants; unit: Participants]
  Had No Concomitant Hypertension | 6764
  Had Concomitant Hypertension | 11485
Concomitant Hyperlipidemia [Count of Participants; unit: Participants]
  Had No Concomitant Hyperlipidemia | 7303
  Had Concomitant Hyperlipidemia | 10946
Concomitant Hyperuricaemia [Count of Participants; unit: Participants]
  Had No Concomitant Hyperuricaemia | 16614
  Had Concomitant Hyperuricaemia | 1635
Concomitant Hepatic Disorder [Count of Participants; unit: Participants]
  Had No Concomitant Hepatic Disorder | 16266
  Had Concomitant Hepatic Disorder | 1983
Concomitant Renal Disorder [Count of Participants; unit: Participants]
  Had No Concomitant Renal Disorder | 16572
  Had Concomitant Renal Disorder | 1677
Concomitant Cardiac Disease [Count of Participants; unit: Participants]
  Had No Concomitant Cardiac Disease | 16032
  Had Concomitant Cardiac Disease | 2217
Concomitant Heart Failure [Count of Participants; unit: Participants]
  Had No Concomitant Heart Failure | 17709
  Had Concomitant Heart Failure | 540
New York Heart Association (NYHA) Heart Failure Classification [Count of Participants; unit: Participants] — NYHA functional classification ranges from Class I (participants with cardiac disease but without resulting limitations of physical activity), Class II (participants with cardiac disease resulting in slight limitation of physical activity), Class III (participants with cardiac disease resulting in marked limitation of physical activity), Class IV (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). Population: This baseline characteristic was analyzed only for participants who had complications of heart failure.
  Participants
    number analyzed (Participants) | 540
    Class I | 354
    Class II | 143
    Class III | 26
    Class IV | 7
    Unknown | 10
Concomitant Stroke-Related Disease [Count of Participants; unit: Participants]
  Had No Concomitant Stroke-Related Disease | 17072
  Had Concomitant Stroke-Related Disease | 1177
Concomitant Allergic Condition [Count of Participants; unit: Participants]
  Had No Concomitant Allergic Condition | 17224
  Had Concomitant Allergic Condition | 1025
Concomitant Malignant Tumor [Count of Participants; unit: Participants]
  Had No Concomitant Malignant Tumor | 17832
  Had Concomitant Malignant Tumor | 417
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 14497
    Had Medical History | 2080
    Unknown | 1672
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 15551
    Had Predisposition to Hypersensitivity | 795
    Unknown | 1903
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 5440
    No | 9156
    Unknown | 3653
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 8089
  Current Smoker | 2330
  Ex-Smoker | 3326
  Unknown | 4504
Hemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP) Value] [Mean (Standard Deviation); unit: Percentage of HbA1c] — Population: The number analyzed is the number of participants with data available for analysis.
  Percentage of HbA1c
    number analyzed (Participants) | 17874
    (all) | 6.88 (0.591)
Dietary Instruction [Count of Participants; unit: Participants] — Reported data was number of participants who received dietary instruction from health care professional at the start of this study as routine medical care.
  Participants
    Instructed | 15433
    Not Instructed | 2816
Exercise Instruction [Count of Participants; unit: Participants] — Reported data was number of participants who received exercise instruction from health care professional at the start of this study as routine medical care.
  Participants
    Instructed | 13909
    Not Instructed | 4340

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Events
Time Frame: Up to Month 36
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Alogliptin 25 mg
Number analyzed (Participants) | 18249
Percentage of Participants | 10.54

2. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at final assessment point (up to Month 36) relative to baseline.
Time Frame: Baseline, and final assessment point (up to Month 36)
Population: The efficacy assessment population was defined as participants who completed the study and had available efficacy data at baseline and post baseline. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Alogliptin 25 mg
Number analyzed (Participants) | 16022
Percent HbA1c | -0.14 (0.777)

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Description: The change in the value of fasting blood glucose level collected at final assessment point (up to Month 36) relative to baseline.
Time Frame: Baseline, and final assessment point (up to Month 36)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligram (mg)/ deciliter (dL)
Arm/Group | Alogliptin 25 mg
Number analyzed (Participants) | 6031
Milligram (mg)/ deciliter (dL) | -5.8 (34.33)

ADVERSE EVENTS:
Time Frame: Up to Month 36
Description: At each visit the investigator had to document any occurrence of adverse events (AEs) and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions (ADRs) were collected and reported on safety results sections here. ADRs are AEs which are in the investigator's opinion of causal relationship to the study treatment..
Arm/Group | Alogliptin 25 mg
All-Cause Mortality (participants affected / at risk) | 20/18249
Serious Adverse Events (participants affected / at risk) | 65/18249
Other Adverse Events (participants affected / at risk) | 41/18249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg (N=18249)
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Marasmus (Metabolism and nutrition disorders) | 1
Completed suicide (Psychiatric disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Depression (Psychiatric disorders) | 1
Cerebellar haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Subdural hygroma (Nervous system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 3
Cholangitis (Hepatobiliary disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 2
Death (General disorders) | 3 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Pyrexia (General disorders) | 1
Sudden death (General disorders) | 5 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
C-reactive protein increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg (N=18249)
Hypoglycaemia (Metabolism and nutrition disorders) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT01964963/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT01964963/SAP_002.pdf